CLINICAL TRIAL: NCT04631107
Title: Phase 2 Randomized Double-Blind Placebo-Controlled 3-Period Single-Dose Crossover Study to Evaluate the Safety and Efficacy of Two Doses of AD-109 in Mild to Moderate Obstructive Sleep Apnea
Brief Title: AD109 Dose Finding in Mild to Moderate OSA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Apnimed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APC-004
Record Dates: First submitted 2020-11-06; First posted 2020-11-17 (Actual); Results first posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-11

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Sequence ABC (Other): AD109 Dose 1- 75 mg (A), then AD109 Dose 2- 37.5 mg (B), then Placebo (C).
  Interventions: Drug: AD109 dose1- A; Drug: AD109 dose2- B; Drug: Placebo- C
- Sequence ACB (Other): AD109 Dose 1- 75 mg (A), then Placebo (C) then AD109 Dose 2- 37.5 mg (B)
  Interventions: Drug: AD109 dose1- A; Drug: AD109 dose2- B; Drug: Placebo- C
- Sequence BAC (Other): AD109 Dose 2- 37.5 mg (B), then AD109 Dose 1- 75 mg (A), then Placebo (C)
  Interventions: Drug: AD109 dose1- A; Drug: AD109 dose2- B; Drug: Placebo- C
- Sequence BCA (Other): AD109 Dose 2- 37.5 mg (B), then Placebo (C), then AD109 Dose 1- 75 mg (A)
  Interventions: Drug: AD109 dose1- A; Drug: AD109 dose2- B; Drug: Placebo- C
- Sequence CAB (Other): Placebo (C), then AD109 Dose 1- 75 mg (A), then AD109 Dose 2- 37.5 mg (B)
  Interventions: Drug: AD109 dose1- A; Drug: AD109 dose2- B; Drug: Placebo- C
- Sequence CBA (Other): Placebo (C), then AD109 Dose 2- 37.5 mg (B), then AD109 Dose 1- 75 mg (A)
  Interventions: Drug: AD109 dose1- A; Drug: AD109 dose2- B; Drug: Placebo- C

INTERVENTIONS:
Drug: AD109 dose1- A — Oral administration at bedtime
  Other Names: AD109 75
Drug: AD109 dose2- B — Oral administration at bedtime
  Other Names: AD109 37.5
Drug: Placebo- C — Oral administration at bedtime

SUMMARY:
This is a randomized, 3-period, placebo-controlled, crossover, phase 2 clinical study to examine the efficacy and safety of 2 doses of AD109 vs placebo in patients with mild obstructive sleep apnea.

DETAILED DESCRIPTION:
Participants underwent initial pre-screening to determine potential study eligibility. Participants selected for further screening had either a previous history of OSA of a severity consistent with enrollment criteria or were at high risk (e.g. as assessed by STOP-Bang Questionnaire score). Only participants who met all non polysomnography (PSG) enrollment criteria at Visit 1 were eligible for a screening PSG.

ELIGIBILITY:
Inclusion Criteria:

* AHI between 5 and 20 events/h
* PGI-S equal to or higher than 1, or one or more of the following symptoms:

  * Snoring or nightime gasping/choking
  * Daytime sleepiness, fatigue or decreased concentration
  * Nonrefreshing sleep, sleep fragmentation (including from nocturia), or morning headache
  * Irritability, decreased mood or libido

Exclusion Criteria:

* History of narcolepsy.
* Clinically significant craniofacial malformation.
* Clinically significant cardiac disease (e.g. rhythm disturbances, coronary artery disease or heart failure or hypertension requiring more than 2 medications for control).
* CPAP should not be used for at least 2 weeks prior to the study
* History of using oral or nasal devices for the treatment of OSA may enroll as long as the devices are not used during participation in the study.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-12-22 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ron Farkas, MD, Study Director — Apnimed
Locations (3):
- United States (3):
  - Pacific Research Network, San Diego, California
  - NeuroTrial Research, Atlanta, Georgia
  - Brian Abaluck, LLC, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Rosenberg R, Abaluck B, Thein S. Combination of atomoxetine with the novel antimuscarinic aroxybutynin improves mild to moderate OSA. J Clin Sleep Med. 2022 Dec 1;18(12):2837-2844. doi: 10.5664/jcsm.10250. PMID 35975547

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 65 participants were screened in the study. Thirty-two participants were randomized.
Pre-assignment Details: Participants who met all enrollment criteria were planned to be randomized to receive the following oral experimental treatments, 1 treatment on each of 3 PSG nights, separated by at least a 1 week washout period. One ineligible participant was inadvertently randomized but not treated. Twenty-seven participants completed the study. Four participants were treated but early terminated from the study.
Groups:
- All Participants: There were three periods with treatment assigned in random order. Treatment A-AD109 dose1 75mg, Treatment B- AD109 37.5 mg, and Treatment C- Placebo. Administered orally at bedtime.
Period: First Intervention (1 Night)
Arm/Group | All Participants
Started | 32
Treatment A | 11
Treatment B | 9
Treatment C | 11
Completed | 31
Not Completed | 1
Not completed — ineligible participant was inadvertently randomized but not treated | 1
Period: Washout 1 Week
Arm/Group | All Participants
Started | 31
Completed | 31
Not Completed | 0
Period: Second Intervention (1 Night)
Arm/Group | All Participants
Started | 31
Treatment A | 11
Treatment B | 9
Treatment C | 9
Completed | 29
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Period: Washout-1 Week
Arm/Group | All Participants
Started | 29
Completed | 29
Not Completed | 0
Period: Third Intervention (1 Night)
Arm/Group | All Participants
Started | 29
Treatment A | 8
Treatment B | 10
Treatment C | 9
Completed | 27
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Groups:
- All Participants: AD109 dose1 75mg, AD109 Dose 2 37.5 mg, and Placebo: Oral administration at bedtime, randomly sequence of all three study products.
Arm/Group | All Participants
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 22
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 31
Hypoxic Burden (HB) [Median (Full Range); unit: (%*min)/hour] — Hypoxic burden is a measure of the overall burden of de-oxygenation (hypoxia) due to upper airway obstructive events for every hour of sleep, measured from the SaO2 signal on the polysomnography done overnight.
  (%*min)/hour | 11.8 [2.08 to 87.78]

OUTCOME MEASURES:

1. Primary Outcome: Change in Hypoxic Burden (HB) Log Transformed - Log10HB[(%*Min)/h]
Description: Change in Hypoxic Burden (HB) is calculated as the oxygen desaturation 'area under the curve' in association with individual apneas and hypopneas. Due to the known logarithmic distribution of HB, data are primarily expressed and analyzed as Log10HB 4%[% min/h]. Raw measurement of HB (%min/h) is defined as the sum of individual areas (%min) divided by total sleep time (h). Events with 4% or greater desaturations were included in the calculation of HB.
Time Frame: 1 night (8 hours)
Measure: Mean (95% Confidence Interval); unit: difference in log10HB[(%*min)/h]
Groups:
- AD109 dose1 vs Placebo: AD109 dose1 75mg: Oral administration at bedtime
- AD109 dose2 vs Placebo: AD109 dose2 37.5mg: Oral administration at bedtime
- Dose 2 vs Dose 1: Low Dose AD109 Versus High Dose AD109
Arm/Group | AD109 dose1 vs Placebo | AD109 dose2 vs Placebo | Dose 2 vs Dose 1
Number analyzed (Participants) | 27 | 27 | 27
difference in log10HB[(%*min)/h] | -0.40 [-0.54 to -0.25] | -0.21 [-0.36 to -0.07] | 0.18 [0.04 to 0.33]

2. Primary Outcome: Change in Hypoxic Burden (HB) Raw Values - HB[(%*Min)/h]
Description: Change in Hypoxic Burden (HB) is calculated as the oxygen desaturation 'area under the curve' in association with individual apneas and hypopneas.
  Raw measurement of HB (%min/h) is defined as the sum of individual areas (%min) divided by total sleep time (h). Events with 4% or greater desaturations were included in the calculation of HB.
Time Frame: 1 night (8 hours)
Measure: Mean (95% Confidence Interval); unit: (%*min)/h
Arm/Group | AD109 dose1 vs Placebo | AD109 dose2 vs Placebo | Dose 2 vs Dose 1
Number analyzed (Participants) | 27 | 27 | 27
(%*min)/h | -6.90 [-10.20 to -3.60] | -4.70 [-8.01 to -1.38] | 2.20 [-1.23 to 5.36]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected for each subject for up to 12 weeks. The overall study duration was up to 12 weeks (Screening period, up to 4 weeks; 3-period crossover, up to 6 weeks; End of Study Evaluation, 2 weeks post crossover period).
Description: The definition of adverse events is the same as clinicaltrials.gov. All AE and SAE were collected from the signing of the informed consent form (ICF) until the end of the study at the timepoints specified in the schedule of assessments
Groups:
- AD109 dose1: AD109 dose1 75mg: Oral administration at bedtime
- AD109 dose2: AD109 dose2 37.5mg: Oral administration at bedtime
- Placebo: Placebo: Oral administration at bedtime
Arm/Group | AD109 dose1 | AD109 dose2 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/28 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/28 | 0/29
Other Adverse Events (participants affected / at risk) | 4/30 | 2/28 | 2/29
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AD109 dose1 (N=30) | AD109 dose2 (N=28) | Placebo (N=29)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Thirst (General disorders) | 0 (0) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-01-06): https://cdn.clinicaltrials.gov/large-docs/07/NCT04631107/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-11): https://cdn.clinicaltrials.gov/large-docs/07/NCT04631107/SAP_001.pdf